CLINICAL TRIAL: NCT05466188
Title: Prediction of Intrahospital Cardiac Arrest Outcomes
Acronym: PREDIHCA
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PREDIHCA
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Outcome CPC Positive: Outcome CPC Positive
  Interventions: Diagnostic Test: CPC
- Outcome CPC Negative: Outcome CPC Negative
  Interventions: Diagnostic Test: CPC

INTERVENTIONS:
Diagnostic Test: CPC — CPC

SUMMARY:
Intrahospital cardiovascular arrest is one of the most common causes of death in hospitalized patients. In contrast to extramural cases of cardiovascular arrest, hospitalized patients often have severe medical conditions that can affect the outcome of resuscitation. Nevertheless, survival rates from resuscitation are better in hospitals than outside, because there is often a rapid start of resuscitation measures and predefined resuscitation standards. Regular CPR training and the availability of defibrillators in all bedside units can also positively influence outcome. Despite these many efforts, survival rates, especially of patients with good neurological outcome, remained stable at low levels even within hospitals in recent years and did not improve.

Most outcome parameters are nowadays well known. (e.g., initial rhythm, age, early defibrillation, etc.) Nevertheless, we still do not know today how relevant the corresponding factors actually are, especially in relation to each other. One approach to this might be machine learning methods such as "random forest", which might be able to create a predictive model. However, this has not been attempted to date.

The hypothesis of this work is to find out if it is possible to accurately predict the probability of surviving an in-hospital resuscitation using the machine learning method "random forest" and if particularly relevant outcome parameters can be identified.

Design: retrospective data analysis of all data sets recorded in the resuscitation register of Kepler University Hospital.

Measures and Procedure: Review of the registry for missing data as well as false alarms of the CPR team and, if necessary, exclusion of these data sets; evaluation of the data sets using the machine learning method random forest.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients suffering cardiac arrest and having been resuscitated by the medical emergency team of the Kepler University Hospital, Linz, Austria in the period of 2006-01-01 to 2018-10-31.

Exclusion Criteria:

* None.

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As described in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 668 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
AUROC for Classification of Outcome CPC | 2006-01-01 to 2018-12-31
  AUROC for Classification of Outcome CPC

SECONDARY OUTCOMES:
Confusion Matrix | 2006-01-01 to 2018-12-31
  Confusion Matrix Results: true positives, true negatives, false positive, false negatives and values calculated from these results.
Descriptive Statistics | 2006-01-01 to 2018-12-31
  Descriptive Statistics (age in years, delay in seconds, gender as male/female, agonal breathing/initial rhythm/airway management/iv-access/witnessed cardiac arrest/use of AED/chest compressions as binary features)
  This outcome measure will compare the individual feature (e. g. height in cm) in one group vs. the other. Significant difference will be described by p-value.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tschoellitsch, MD, Principal Investigator — Kepler University Hospital and Johannes Kepler University, Linz, Austria
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No